CLINICAL TRIAL: NCT05968703
Title: Neurostimulation of the Nucleus Basalis of Meynert for the Cognitive-Motor Syndrome in Parkinson's Disease
Brief Title: Combined STN and NBM Deep Brain Stimulation for Mild Cognitive Impairment in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helen M. Bronte-Stewart (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Helen M. Bronte-Stewart, Professor of Neurology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70608; UG3NS128150 (NIH); UH3NS128150 (NIH)
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: deep brain stimulation; cognition; DBS; parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All participants will receive the interventional treatment. Two different surgical trajectories will be used for placing the leads in the NBM. Half the cohort will be randomized to each trajectory.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vertical Nuclear Trajectory (Experimental): Participants will receive combined STN + NBM DBS. The lead placed within the NBM will use a vertical trajectory targeting the nucleus itself.
  Interventions: Device: Combined STN+NBM DBS
- Lateral NBM Bundle Trajectory (Experimental): Participants will receive combined STN + NBM DBS. The lead placed within the NBM will use a lateral trajectory targeting the lateral efferent bundle from the NBM
  Interventions: Device: Combined STN+NBM DBS

INTERVENTIONS:
Device: Combined STN+NBM DBS — This intervention is a 4-lead deep brain stimulation approach targeting the Subthalamic Nucleus (STN) and Nucleus Basalis of Meynert (NBM)

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of a novel deep brain stimulation (DBS) of the Subthalamic Nucleus (STN) and Nucleus Basalis of Meynert (NBM) to treat cognitive and cognitive-motor symptoms in individuals with Parkinson's disease. The main question it aims to answer is:

Is a combined deep brain stimulation approach targeting the STN and NBM with four DBS leads safe and tolerable for cognitive and cognitive-motor symptoms in individuals with Parkinson's disease with Mild Cognitive Impairment. Ten participants are anticipated to be enrolled.

Participants will undergo a modification of the traditional STN DBS approach for motor symptoms of PD. In addition to the two leads placed within the STN, two additional leads will be placed with the NBM for treatment of cognitive and cognitive-motor symptoms. Novel stimulation patterns will be used within the NBM to target cognitive and cognitive-motor symptoms using an investigational software. Participants will be followed over two years while receiving this therapy with assessments at baseline and every six months. Assessments will include a combination of neuropsychological evaluations, cognitive assessments, motor tasks (including gait/walking), and questionnaires to evaluate the treatment. Two different surgical trajectories will be used, with half the cohort randomized to each group. This will allow comparison of the impact of surgical trajectory on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (PD)
* Approved (or planning on) for subthalamic nucleus (STN) deep brain stimulation (DBS)
* Willingness to withdraw from clinical medication regimen when necessary for research visits
* Ability to provide informed consent

Exclusion Criteria:

* Dementia
* Unstable medical, psychiatric conditions including significant untreated depression, history of suicidal attempt, or current suicide ideation
* History of seizures
* Pregnant
* Requires MRI
* Unable to walk 100 feet without an assistive device

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From baseline to 1 year into treatment
  Any untoward medical occurrence that occurs during this study whether or not considered related to the study device, study procedures, or study requirements that is identified or worsens during the duration of the study
Swing Time Coefficient of Variation | From baseline to 1 year into treatment
  Swing time variability will be measured using the dual force plates in the SIP task and IMUs for TBC. It is defined as the mean swing time coefficient of variation (CV) of both legs.

SECONDARY OUTCOMES:
Percent Time Freezing | From baseline to 1 year into treatment
  Duration of freezing episodes during SIP will be measured using IMUs and force plates using a validated offline algorithm.
Stride Time Coefficient of Variation | From baseline to 1 year into treatment
  Stride time coefficient of variation will be measured using the dual force plates in the SIP task and IMUs. Stride time coefficient of variation is defined as the mean stride time coefficient of variation (CV) of both legs. A greater stride time CV is indicative of less rhythmic gait/stepping.
Shank Angular Velocity | From baseline to 1 year into treatment
  Shank angular velocity will be measured from IMUs work on the participant's leg/ankle. Reductions in this value are indicative of FOG and gait impairment.
Tapping Speed | From baseline to 1 year into treatment
  The interstrike-interval of alternating tapping will be measured using an engineered piano keyboard. A higher interstrike-interval indicates slower tapping
Tapping Rhythmicity | From baseline to 1 year into treatment
  The variability of the interstrike-interval of alternating tapping, as quantified by the coefficient of variation, will be measured using an engineered piano keyboard. A higher coefficient of variation indicates worse rhythmicity
MDS-UPDRS III Score | From baseline to 1 year into treatment
  PD symptoms will be assessed clinically using the MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Section III. This is a motor examination to evaluate speech, facial expression, tremor at rest, action or postural tremor of hands, rigidity, finger taps, hand movements, rapid alternating movement of hands, leg agility, arising from chair, posture, gait, freezing of gait, posture, body bradykinesia, and postural stability. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 132.
SAT Score | From baseline to 1 year into treatment
  Each trial of the SAT will be categorized as a Hit (H), Miss (M), or False Alarm (FA). The SAT score is defined as ((H - FA) / [2× (H + FA) - (H + FA)2]), which ranges from - 1.0 (100% incorrect performance; all misses and false alarms) to +1.0 (100% correct performance; all hits and correct rejections).
Percent False Positives | From baseline to 1 year into treatment
  The percent of false positives during the SAT.
Percent Misses | From baseline to 1 year into treatment
  The percent of misses of total trials during the SAT
Average + standard deviation of response time | From baseline to 1 year into treatment
  The average and standard deviation of the response time during the SAT.
Goal-directed focus of attention | From baseline to 1 year into treatment
  Hit rate during the first minute in the no- distractor condition for the CTET.
Sustained attention | From baseline to 1 year into treatment
  Hit rate change slope in no-distractor condition for the CTET.
Distractibility | From baseline to 1 year into treatment
  Hit rate difference between no-distractor and distractor conditions for the CTET.
Parkinson's Disease - Cognitive Rating Scale (PD-CRS) | From baseline to 1 year into treatment
  Cognitive scale composed of 9 tasks that assesses the full range of cognitive dysfunction in PD. It is a scale of 0 to 134, with 134 being the best score.
Montreal Cognitive Assessment (MoCA) | From baseline to 1 year into treatment
  Total score to assess of this rapid screening test of different cognitive domains. It is a scale of 0 to 30, with 30 being the best score.
Trails A | From baseline to 1 year into treatment
  The time it takes to complete the task and errors.
Trails B | From baseline to 1 year into treatment
  The time it takes to complete the task and errors.
Symbol Digit Modalities (SDMT) Oral and Written | From baseline to 1 year into treatment
  The summation of the number of correct substitutions within the 90 second interval.
visual puzzles from the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | From baseline to 1 year into treatment
  Percentile of performance on visual puzzles for participant's demographic.
Judgement of Line Orientation | From baseline to 1 year into treatment
  Percentile of performance on judgement of line orientation for participant's demographic.
Patient Health Questionnaire-9 (PHQ-9) | From baseline to 1 year into treatment
  Total score on questionnaire regarding participant's mood the last 2 weeks. The scale ranges from 0 to 27 with a score of 27 indicating the most severe symptoms.
General Anxiety Disorder-7 (GAD-7) | From baseline to 1 year into treatment
  Total score on questionnaire regarding participant's anxiety the last two weeks.The scale ranges from 0 to 21 with a score of 21 indicating the most severe symptoms.
MDS-UPDRS I | From baseline to 1 year into treatment
  Total score evaluating the non-motor aspects of experiences of daily living. It is a scale from 0 to 52 with 52 being the most severe symptoms.
MDS-UPDRS II | From baseline to 1 year into treatment
  Total score evaluating the motor aspects of experiences of daily living. It is a scale from 0 to 52 with 52 being the most severe symptoms.
MDS-UPDRS IV | From baseline to 1 year into treatment
  Total score of motor complications experienced by the participant. It is a scale from 0 to 24 with 24 being the most severe symptoms.
Neuropsychiatric Inventory (NPI) | From baseline to 1 year into treatment
  Total score for symptom severity and distress via questionnaire. It is a scale from 0 to 60 with 60 indicating worse symptoms.
Parkinson's Disease Questionnaire-39 (PDQ-39) | From baseline to 1 year into treatment
  Total score for Parkinson's disease-specific health related quality over the last month across 8 quality of life dimensions assessed via questionnaire. Score ranges from 0 to 100 with 100 indicating more symptoms and problems.
Caregiver Burden Assessment | From baseline to 1 year into treatment
  Total score on caregiver self-report to assess the stress-levels of family caregivers. It is a scale from 0 to 88 with higher scores indicating greater or worse burden.

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Bronte-Stewart, MD MSE, Principal Investigator — Stanford University
Locations (1):
- Stanford Neuroscience Health Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded to the Data Archive for the BRAIN Initiative (DABI).
Supporting Information: CSR
Time Frame: The IPD is anticipated to be available in approximately three months after study completion
Access Criteria: DABI is openly available